CLINICAL TRIAL: NCT01834079
Title: Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Optic Nerve Disease. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Study the Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Optic Nerve Disease
Acronym: OND
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00104
Record Dates: First submitted 2013-02-26; First posted 2013-04-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Optic Atrophy
Keywords: Optic Atrophy,Stem cell therapy
MeSH Terms: conditions — Optic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STEM CELL (Other): intra thecal injection of MNC stem cell therapy
  Interventions: Biological: STEM CELL THERAPY

INTERVENTIONS:
Biological: STEM CELL THERAPY — Autologous stem cells(MNCs ) intra thecal .Intra thecal transplantation of single arm autologous MNCs 100 millions per dose in 3 divided doses at interval of 7 days,Intrathecal/Intravenous .Follow up will be taken to three Months or as required
  Other Names: Intrathecal transplantation of autologous stem cells

SUMMARY:
This is a Single arm, Single centre trial to check the safety and efficacy of bone marrow derived autologous mono nuclear cell(100 millions per dose )clinical trial to be conducted for 36 months in patients with optic nerve diseases.

DETAILED DESCRIPTION:
Optic Nerve Diseases: Conditions which produce injury or dysfunction of the second cranial or optic nerve, which is generally considered a component of the central nervous system. Damage to optic nerve fibres may occur at or near their origin in the retina, at the optic disk, or in the nerve, optic chiasm, optic tract, or lateral geniculate nuclei. Clinical manifestations may include decreased visual acuity and contrast sensitivity, impaired color vision, and an afferent papillary defect. primary out put of clinical study is to measures Improvement in visual loss and improvement in idiopathic intra cranial.This is a Single arm, Single centre trial to check the safety and efficacy of bone marrow derived autologous mono nuclear cell(100 millions per dose )clinical trial to be conducted for 36 months .

ELIGIBILITY:
Inclusion Criteria:

* Patient Should suffer from Optic Nerve diseases Like Diabetic Retinopathy, retinal pigmentation
* age in between 18 to 50
* Willingness to undergo Bone Marrow derived autologous cell therapy.
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the require Informed consent form(ICF) for the study.
* A ability and willingness to regular visit to hospital for protocol and follow up.

Exclusion Criteria:

* Patients with pre - existing or Current systemic disease such as lung , liver ( exception; History of uncomplicated Hepatitis A),gastrointestinal, Cardiac , Immunodeficiency,(including HIV) Or laboratory Investigation that could cause a neurological defect including Syphilis, clinically relevant polyneuropathy) etc.
* History of Life threatening Allergic or immune- mediated reaction
* Haemodynamically Unstable.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in degeneration of the Optic nerve with improvement in vision | 6 Months

SECONDARY OUTCOMES:
Increase in Visual Function | 6 months
Improvement in idiopathic intra cranial hypertension | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India